CLINICAL TRIAL: NCT06717347
Title: A Randomized, Open-Label, Multicenter, Phase 3 Study of Zilovertamab Vedotin (MK-2140) in Combination With R-CHP Versus R-CHOP in Participants With Previously Untreated Diffuse Large B-Cell Lymphoma (DLBCL) (waveLINE-010)
Brief Title: A Study to Evaluate Zilovertamab Vedotin (MK-2140) Combination With Rituximab Plus Cyclophosphamide, Doxorubicin, and Prednisone (R-CHP) Versus Rituximab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Participants With Previously Untreated DLBCL (MK-2140-010)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2140-010; MK-2140-010 (Other: MSD); 2024-515566-13-00 (Registry Identifier: EU CT); U1111-1309-3971 (Registry Identifier: UTN); jRCT2061240099 (Other: jRCT)
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Prednisolone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zilovertamab vedotin + Rituximab + Cyclophosphamide, Doxorubicin, Prednisone (R-CHP) (Experimental): Participants receive a dose of zilovertamab vedotin (1.75 mg/kg) plus 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar administered by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 6 cycles (up to approximately 4 months) plus 2 cycles of rituximab or biosimilar for participants with high risk DLBCL. Participants also receive 100 mg prednisone or prednisolone via oral tablet per day during Days 1-5 of each 21-day cycle for up to 6 cycles (up to approximately 4 months).
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone; Drug: Rescue medication
- Rituximab + Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (R-CHOP) (Active Comparator): Participants receive 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar, 1.4 mg/m^2 vincristine administered by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 6 cycles (up to approximately 4 months) plus 2 cycles of rituximab or biosimilar for participants with high risk DLBCL. Participants also receive 100 mg prednisone or prednisolone via oral tablet per day during Days 1-5 of each 21-day cycle for up to 6 cycles (up to approximately 4 months).
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone; Drug: Vincristine

INTERVENTIONS:
Biological: Zilovertamab vedotin — IV infusion
  Other Names: MK-2140; VLS-101
  Arms: Zilovertamab vedotin + Rituximab + Cyclophosphamide, Doxorubicin, Prednisone (R-CHP)
Biological: Rituximab — IV infusion
  Other Names: RITUXAN®
Drug: Cyclophosphamide — IV infusion
  Other Names: CYTOXAN®; NEOSAR®
Drug: Doxorubicin — IV infusion
  Other Names: ADRIAMYCIN®
Biological: Rituximab Biosimilar — IV infusion
  Other Names: TRUXIMA®; RUXIENCE®; RIABNI®
Drug: Prednisone — Per Approved Product Label
Drug: Prednisolone — Oral administration
Drug: Vincristine — IV infusion
  Arms: Rituximab + Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (R-CHOP)
Drug: Rescue medication — Participants receive rescue medication at the investigator's discretion, per approved product label. The recommended rescue medication is granulocyte colony-stimulating factor (G-CSF).
  Arms: Zilovertamab vedotin + Rituximab + Cyclophosphamide, Doxorubicin, Prednisone (R-CHP)

SUMMARY:
The purpose of this study is to evaluate if zilovertamab vedotin with standard treatment can help people live longer without the cancer growing or spreading than people who receive standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL), by prior biopsy, based on local testing according to the WHO classification of neoplasms of the hematopoietic and lymphoid tissues
* Has positron emission tomography (PET) positive disease at screening, defined as 4 to 5 on the Lugano 5-point scale
* Has received no prior treatment for their DLBCL
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 assessed within 7 days before randomization
* Has an ejection fraction ≥45% as determined by either echocardiogram (ECHO) or multigated acquisition (MUGA)
* Human immunodeficiency virus (HIV) infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy and have undetectable HBV viral load prior to randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

* Has a history of transformation of indolent disease to DLBCL
* Has received a diagnosis of primary mediastinal B-cell lymphoma (PMBCL) or Grey zone lymphoma
* Has Ann Arbor Stage I DLBCL
* Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication
* Has clinically significant pericardial or pleural effusion
* Has ongoing Grade >1 peripheral neuropathy
* Has a demyelinating form of Charcot-Marie-Tooth disease
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has ongoing corticosteroid therapy
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Known additional malignancy that is progressing or has required active treatment within the past 2 years
* Known active central nervous system (CNS) lymphoma
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has active infection requiring systemic therapy
* Has concurrent active HBV (defined as HBsAg positive and detectable HBV DNA) and HCV (defined as anti-HCV antibody positive and detectable HCV ribonucleic acid (RNA)) infection
* Has history of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2029-07-02 (Estimated); Study Completion 2032-03-29 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to ~ 50 months
  PFS is defined as the time from randomization to the first documented disease progression per Lugano response criteria by blinded independent central review (BICR) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Complete Response at End of Treatment (CR at EOT) | Up to ~ 32 months
  CR at EOT is defined as a CR per Lugano response criteria as assessed by BICR at end of treatment. Participants with missing data or who discontinue treatment or study prior to reaching EOT will be considered non-responders and included in the total number of participants.
Overall Survival (OS) | Up to ~ 74 months
  OS is defined as the time from randomization to death due to any cause.
Event-free Survival (EFS) | Up to ~ 74 months
  EFS is defined as the time from randomization to any of the following events: progressive disease that precludes surgery, local or distant recurrence, second primary malignancy or death due to any cause. The EFS for all participants will be presented.
Duration of Complete Response (DurCR) | Up to ~ 74 months
  For participants who demonstrate CR at EOT per Lugano response criteria by BICR, duration of complete response is defined as the time from the first documented evidence of CR at or before EOT until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~ 9 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to ~ 6 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Change From Baseline in Health-Related Quality Of Life (HRQoL) on Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Trial Outcome Index (TOI) Score | Baseline and Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on FACT-Lym Total Score | Baseline and Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on FACT-Lym Physical Wellbeing (PWB) Score | Baseline and Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) Neurotoxicity Subscale Score | Baseline and Week 25
  The FACT GOG-NTX provides a targeted assessment of symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity. It is an 11-item questionnaire designed to measure the neurotoxicity subscale. The scoring of FACT GOG-NTX is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. To produce a Neurotoxicity Subscale score (range 0-44), multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (236):
- United States (27):
  - The University of Arizona Cancer Center - North Campus ( Site 0124), Tucson, Arizona
  - Cancer Blood and Specialty Clinic ( Site 0109), Los Alamitos, California
  - Cedars-Sinai Medical Center ( Site 0115), Los Angeles, California
  - Pacific Hematology Oncology Associates ( Site 0131), San Francisco, California
  - Bioresearch Partner ( Site 0157), Hialeah, Florida
  - Orlando Health Cancer Institute ( Site 0169), Ocoee, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0172), Orange City, Florida
  - Cancer Care Specialists of Illinois ( Site 0152), O'Fallon, Illinois
  - Fort Wayne Medical Oncology and Hematology ( Site 0149), Fort Wayne, Indiana
  - Cotton O'Neil Cancer Center ( Site 0108), Topeka, Kansas
  - University of Kentucky ( Site 0106), Lexington, Kentucky
  - Norton Women's and Children's Hospital-Norton Cancer Institute - St. Matthews ( Site 0163), Louisville, Kentucky
  - Corewell Health ( Site 0130), Grand Rapids, Michigan
  - Circuit Clinical - SSM Health Cancer Care DePaul ( Site 0166), Bridgeton, Missouri
  - Truman Medical Center ( Site 0122), Kansas City, Missouri
  - OptumCare Cancer Care ( Site 0121), Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada ( Site 0113), Las Vegas, Nevada
  - New York Oncology Hematology, P.C. ( Site 0129), Albany, New York
  - Prisma Health - Upstate ( Site 0158), Greenville, South Carolina
  - Sanford Cancer Center ( Site 0143), Sioux Falls, South Dakota
  - The University of Tennessee Medical Center ( Site 0142), Knoxville, Tennessee
  - Center for Oncology and Blood Disorders ( Site 0153), Houston, Texas
  - Houston Methodist Cancer Center ( Site 0154), Houston, Texas
  - University of Virginia Cancer Center ( Site 0138), Charlottesville, Virginia
  - Virginia Cancer Institute ( Site 0148), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0132), Roanoke, Virginia
  - SSM Health Dean Medical Group ( Site 0140), Madison, Wisconsin
- Argentina (8):
  - Clinica Adventista Belgrano ( Site 0309), Caba., Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0306), Mar del Plata, Buenos Aires
  - Hospital Universitario Austral ( Site 0307), Pilar, Buenos Aires
  - Hospital Aleman ( Site 0301), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 0311), Rosario, Santa Fe Province
  - C.I.C.E. 9 de Julio ( Site 0305), San Miguel de Tucumán, Tucumán Province
  - Hospital Italiano de Buenos Aires ( Site 0304), CABA
  - Clinica EL Castaño ( Site 0312), San Juan
- Australia (5):
  - Townsville University Hospital ( Site 3006), Douglas, Queensland
  - Royal Adelaide Hospital ( Site 3001), Adelaide, South Australia
  - Grampians Health ( Site 3003), Ballarat, Victoria
  - Northern Hospital ( Site 3002), Melbourne, Victoria
  - Royal Perth Hospital-Haematology ( Site 3004), Perth, Western Australia
- Belgium (2):
  - AZ Sint-Maarten, Campus Leopoldstraat 2 ( Site 1102), Mechelen, Antwerpen
  - ASBL CHU Helora - Hôpital de Mons - Site Kennedy ( Site 1103), Mons, Hainaut
- Brazil (9):
  - CEONC ( Site 0412), Cascavel, Paraná
  - Hospital Erasto Gaertner ( Site 0401), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer ( Site 0407), Natal, Rio Grande do Norte
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina ( Site 0403), Florianópolis, Santa Catarina
  - Hope ( Site 0413), Ribeirão Preto, São Paulo
  - Clinica Advanze ( Site 0411), São Carlos, São Paulo
  - F. F. R. M. São Jose do Rio Preto ( Site 0404), SJRP, São Paulo
  - Hospital Paulistano ( Site 0406), São Paulo
  - Hospital das Clinicas FMUSP ( Site 0402), São Paulo
- Canada (2):
  - Lakeridge Health - The R.S. McLaughlin Durham Regional Cancer Centre (MDRCC) ( Site 0206), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 0204), Toronto, Ontario
- Chile (9):
  - IC La Serena Research ( Site 0504), La Serena, Coquimbo Region
  - Oncocentro Valdivia ( Site 0506), Valdivia, Los Ríos Region
  - Centro de Estudios Clínicos SAGA ( Site 0508), Santiago, Region M. de Santiago
  - FALP ( Site 0501), Santiago, Region M. de Santiago
  - Clinica Inmunocel ( Site 0503), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 0512), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0502), Santiago, Region M. de Santiago
  - Centro de Investigaciones ( Site 0511), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 0510), Concepción, Región del Biobío
- China (24):
  - Anhui Provincial Cancer Hospital ( Site 3124), Hefei, Anhui
  - Peking University Third Hospital ( Site 3102), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3101), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 3113), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital. ( Site 3119), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 3120), Xiamen, Fujian
  - Sun Yat-sen University Cancer Center ( Site 3121), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University ( Site 3122), Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 3123), Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University ( Site 3112), Guiyang, Guizhou
  - Hubei Cancer Hospital ( Site 3125), Wuhan, Hubei
  - Affiliated Hospital of Nantong University ( Site 3117), Nantong, Jiangsu
  - Jiangxi Cancer Hospital ( Site 3118), Nanchang, Jiangxi
  - The First Hospital Of Jilin University ( Site 3103), Changchun, Jilin
  - Shandong Cancer Hospital ( Site 3108), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 3104), Linyi, Shandong
  - Fudan University Shanghai Cancer Center ( Site 3115), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 3106), Taiyuan, Shanxi
  - 1st Affil Hosp of Med College of Xi'an Jiaotong University ( Site 3107), Xi’an, Shanxi
  - Sichuan Cancer Hospital. ( Site 3111), Chengdu, Sichuan
  - West China Hospital, Sichuan University ( Site 3110), Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hosp CAMS&PUMC ( Site 3105), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital ( Site 3109), Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang Medical University ( Site 3116), Hangzhou, Zhejiang
- Colombia (5):
  - Hospital Pablo Tobon Uribe ( Site 0604), Medellín, Antioquia
  - Hospital Universitario San Ignacio ( Site 0607), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0603), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0601), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 0602), Cali, Valle del Cauca Department
- Denmark (2):
  - Regionshospitalet Gødstrup ( Site 1301), Herning, Central Jutland
  - Aalborg University Hospital ( Site 1302), Aalborg, North Denmark
- France (14):
  - Centre Antoine-Lacassagne ( Site 1514), Nice, Alpes-Maritimes
  - Hopital Saint Louis, Centre Hospitalier de La Rochelle ( Site 1511), La Rochelle, Charente-Maritime
  - CHU Dijon Bourgogne ( Site 1516), Dijon, Cote-d Or
  - Institut Curie - site Saint-Cloud ( Site 1501), Saint-Cloud, Hauts-de-Seine
  - CHU GRENOBLE ALPES ( Site 1518), La Tronche, Isere
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren ( Site 1512), Limoges, Limousin
  - Centre Hospitalier Régional Metz Thionville - Hôpital de Mercy ( Site 1515), Metz, Moselle
  - Centre Hospitalier de Dunkerque ( Site 1513), Dunkirk, Nord
  - Centre Hospitalier Universitaire Estaing ( Site 1508), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier de la Cote Basque ( Site 1509), Bayonne, Pyrenees-Atlantiques
  - Centre Henri Becquerel ( Site 1517), Rouen, Seine-Maritime
  - HIA Sainte Anne ( Site 1506), Toulon, Var
  - Centre Hospitalier d'Avignon ( Site 1505), Avignon, Vaucluse
  - CHD Vendee ( Site 1502), La Roche-sur-Yon, Vendee
- Greece (4):
  - Evangelismos General Hospital of Athens ( Site 1602), Athens, Attica
  - General Hospital of Athens "Laiko"-Hematology Department ( Site 1603), Athens, Attica
  - Attikon University General Hospital of Athens ( Site 1604), Athens, Attica
  - University General Hospital of Alexandroupoli ( Site 1601), Alexandroupoli, Evros
- Guatemala (3):
  - MEDI-K ( Site 0701), Guatemala City
  - CELAN,S.A ( Site 0702), Guatemala City
  - Cen Integral Onco Gastro y Hemato Onco Guatemala S.A. ( Site 0703), Guatemala City
- Hong Kong (2):
  - Princess Margaret Hospital ( Site 3202), Hong Kong
  - Queen Mary Hospital ( Site 3201), Hong Kong
- Hungary (3):
  - Debreceni Egyetem Klinikai Kozpont ( Site 1702), Debrecen, Hajdú-Bihar
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház ( Site 1704), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Tolna Vármegyei Balassa János Kórház ( Site 1710), Szekszárd, Tolna County
- Israel (4):
  - Carmel Hospital ( Site 1903), Haifa
  - Hadassah Medical Center ( Site 1901), Jerusalem
  - Sourasky Medical Center ( Site 1904), Tel Aviv
  - Poria Medical Center ( Site 1902), Tiberias
- Italy (11):
  - Fondazione IRCCS San Gerardo dei Tintori ( Site 2008), Monza, Lombardy
  - IRCCS Crob ( Site 2002), Rionero in Vulture, Potenza
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia ( Site 2010), Candiolo, Torino
  - AOU delle Marche Ospedali Riuniti di Ancona ( Site 2011), Ancona
  - Azienda Ospedaliera Spedali Civili di Brescia-Hemathology ( Site 2001), Brescia
  - IRCCS Ospedale San Raffaele ( Site 2012), Milan
  - IEO Istituto Europeo di Oncologia ( Site 2009), Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità ( Site 2004), Novara
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO ( Site 2005), Palermo
  - Ospedale Santa Maria delle Croci ( Site 2006), Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 2003), Roma
- Japan (19):
  - Nagoya University Hospital ( Site 3309), Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center ( Site 3321), Matsuyama, Ehime
  - Kobe City Medical Center General Hospital ( Site 3318), Kobe, Hyōgo
  - Kanazawa University Hospital ( Site 3308), Kanazawa, Ishikawa-ken
  - Tokai University Hospital ( Site 3302), Isehara, Kanagawa
  - Tohoku University Hospital ( Site 3301), Sendai, Miyagi
  - Kindai University Hospital ( Site 3310), Sakai, Osaka
  - Saitama Medical University Hospital ( Site 3305), Iruma-gun, Saitama
  - Juntendo University Hospital ( Site 3307), Bunkyo, Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 3323), Bunkyo, Tokyo
  - University of Yamanashi Hospital ( Site 3320), Chūō, Yamanashi
  - Chiba Cancer Center ( Site 3314), Chiba
  - Kyushu University Hospital ( Site 3313), Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital ( Site 3322), Hiroshima
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 3315), Kyoto
  - University of Miyazaki Hospital ( Site 3319), Miyazaki
  - Okayama University Hospital ( Site 3311), Okayama
  - Osaka Metropolitan University Hospital ( Site 3317), Osaka
  - Yamagata University Hospital ( Site 3312), Yamagata
- Malaysia (5):
  - Queen Elizabeth Hospital ( Site 3405), Kota Kinabalu, Sabah
  - Sarawak General Hospital ( Site 3402), Kuching, Sarawak
  - Hospital Miri ( Site 3403), Miri, Sarawak
  - Sunway Medical Centre ( Site 3406), Petaling Jaya, Selangor
  - Hospital Ampang ( Site 3404), Selangor Darul Ehsan, Selangor
- Mexico (7):
  - CIMAB SA de CV ( Site 0807), Torreón, Coahuila
  - Grupo Ollin Care ( Site 0806), Pachuca, Hidalgo
  - Health Pharma Professional Research S.A. de C.V. ( Site 0801), Mexico City, Mexico City
  - Centro de Infusion Superare ( Site 0804), Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec ( Site 0803), Morelia, Michoacán
  - Hospital Universitario ""Dr. Jose Eleuterio Gonzalez"" ( Site 0802), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0805), Oaxaca City
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis ( Site 2103), Dordrecht, South Holland
  - Meander Medisch Centrum ( Site 2101), Amersfoort, Utrecht
- Peru (5):
  - Clínicas AUNA Sede Chiclayo ( Site 0904), Chiclayo, Lambayeque
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 0901), Surquillo, Muni Metro de Lima
  - Clínica San Felipe ( Site 0906), Lima
  - Hospital Nacional Edgardo Rebagliati Martins ( Site 0903), Lima
  - Hospital Nacional Dos De Mayo ( Site 0905), Lima
- Poland (5):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 2201), Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. J. Korczaka w Słupsku ( Site 2210), Słupsk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2208), Gliwice, Silesian Voivodeship
  - Pratia Onkologia Katowice ( Site 2204), Katowice, Silesian Voivodeship
  - Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji z Warmińsko-Mazurskim Centrum Onko ( Site 2205), Olsztyn, Warmian-Masurian Voivodeship
- Portugal (2):
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 2306), Braga
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E. ( Site 2302), Porto
- Puerto Rico (2):
  - BRCR Global - Mayaguez ( Site 1003), Mayagüez
  - Auxilio Mutuo Cancer Center ( Site 1001), San Juan
- Romania (4):
  - Spitalul Clinic Colțea ( Site 2401), Bucharest, București
  - Institutul Oncologic Cluj ( Site 2404), Cluj-Napoca, Cluj
  - Centrul de Diagnostic si Tratament Oncologic Brasov ( Site 2402), Brasov
  - Spital Judetean Sibiu ( Site 2405), Sibiu
- Singapore (2):
  - National University Hospital ( Site 3702), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 3701), Singapore, Central Singapore
- South Africa (4):
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 2506), Pretoria, Gauteng
  - Netcare Pretoria East Hospital ( Site 2502), Pretoria, Gauteng
  - Haemalife ( Site 2501), Cape Town, Western Cape
  - Groote Schuur Hospital ( Site 2504), Cape Town, Western Cape
- South Korea (7):
  - National Cancer Center- Center for Hemotologic malignancy ( Site 3806), Goyang-si, Kyonggi-do
  - Pusan National University Hospital ( Site 3804), Busan, Pusan-Kwangyokshi
  - Chungnam National University Hospital ( Site 3801), Daejeon, Taejon-Kwangyokshi
  - Severance Hospital, Yonsei University Health System ( Site 3802), Seoul
  - Asan Medical Center ( Site 3803), Seoul
  - Samsung Medical Center ( Site 3807), Seoul
  - St.Mary's H., Youido ( Site 3805), Seoul
- Spain (9):
  - Hospital Universitario Virgen Macarena ( Site 2608), Seville, Andalusia
  - ICO L Hospitalet ( Site 2601), L'Hospitalet de Llobregat, Barcelona
  - H. Insular de Gran Canaria ( Site 2606), Las Palmas de Gran Canaria, Las Palmas
  - Hospital General Universitario Dr. Balmis ( Site 2604), Alicante, Valenciana, Comunitat
  - Hospital del Mar ( Site 2610), Barcelona
  - Hospital General Universitario 12 de Octubre ( Site 2605), Madrid
  - Hospital Universitario La Paz ( Site 2611), Madrid
  - Hospital Virgen de la Victoria ( Site 2609), Málaga
  - Hospital Universitario Miguel Servet ( Site 2607), Zaragoza
- Switzerland (4):
  - Kantonspital Baden ( Site 2703), Baden, Canton of Aargau
  - Cantonal Hospital St.Gallen-Oncology & Hematology ( Site 2702), Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale Bellinzona e Valli ( Site 2701), Bellinzona, Canton Ticino
  - Ospedale Italiano Lugano (OIL) ( Site 2705), Lugano, Canton Ticino
- Taiwan (6):
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 3903), Taoyuan, Taoyuan
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3905), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 3902), Tainan
  - National Taiwan University Hospital ( Site 3901), Taipei
  - Mackay Memorial Hospital ( Site 3908), Taipei
  - Tri-Service General Hospital ( Site 3906), Taipei
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital ( Site 4001), Bangkoknoi, Bangkok
  - Chulalongkorn University ( Site 4003), Pathumwan, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 4002), Muang, Chiang Mai
- Turkey (Türkiye) (8):
  - Ondokuz Mayıs Universitesi ( Site 2806), Korfez Mahallesi, Samsun
  - Namık Kemal University Medical Faculty ( Site 2807), Suleymanpasa, Tekirdas
  - Baskent Universitesi Adana Dr. Turgut Noyan UAM ( Site 2809), Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi ( Site 2803), Ankara
  - Hacettepe Universite Hastaneleri ( Site 2810), Ankara
  - Ankara University Faculty of Medicine ( Site 2801), Ankara
  - Antalya Egitim ve Arastirma Hastanesi ( Site 2805), Antalya
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi ( Site 2804), Istanbul
- Ukraine (8):
  - MNPE ClinCenter of Oncology,Hematology,Transplantology and Palliative Care of CherkasyRegCouncil ( Site 2904), Cherkasy, Cherkasy Oblast
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council" ( Site 2906), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Khmelnytskyi Regional Hospital ( Site 2907), Khmelnytskiy, Khmelnytskyi Oblast
  - Institute of Blood Pathology and Transfusion Medicine AMS Ukraine ( Site 2903), Lviv, Lviv Oblast
  - SNPE National Cancer Institute ( Site 2902), Kyiv
  - Universal Clinic Oberig ( Site 2908), Kyiv
  - SI National Research Center of Radiation Medicine, Hematology, Oncology ( Site 2901), Kyiv
  - Public Non-Profit Enterprise Kyiv City Clinical Hospital #9 under the Executive Body of Kyiv City Co ( Site 2905), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/